CLINICAL TRIAL: NCT04320290
Title: Hepatitis C Viral Kidneys Used for Non-Viremic Recipients
Brief Title: HCV + to HCV - Kidney Transplant
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: New Related Protocol to be submitted
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Nahel Elias, M.D., Surgical Director, Kidney Transplant, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020P000374
Record Dates: First submitted 2020-03-23; First posted 2020-03-24 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Kidney Failure; Hepatitis C
Keywords: Kidney Transplant; Kidney Failure; HCV; Hepatitis C
MeSH Terms: conditions — Renal Insufficiency; Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with Direct Acting Antiviral for HCV (Experimental): 8 weeks of treatment with HCV Direct Acting Antiviral tablet
  Interventions: Drug: Direct Acting Antivirals

INTERVENTIONS:
Drug: Direct Acting Antivirals — 8 weeks of DAA treatment
  Other Names: Direct Acting Antiviral HCV Treatment

SUMMARY:
This is a single center study characterizing the experience of administration of 8 weeks of pan-genotypic DAA therapy in kidney transplantation to prevent the transmission of hepatitis C virus infection from an HCV-positive donor kidney to an HCV-negative recipient.

DETAILED DESCRIPTION:
The goal of this study is to determine if 8 weeks of preemptive and sustained administration of pan-genotypic DAA therapy after kidney transplant prevents the transmission of hepatitis C virus (HCV) infection from an HCV-positive donor kidney to an HCV-naive recipient.

ELIGIBILITY:
Recipient Inclusion Criteria:

* Met MGH transplant center criteria and already listed for kidney transplant
* Must agree to birth control. Women must agree to use birth control in accordance with Mycophenolate Risk Evaluation and Mitigation Strategy and at least one barrier method
* No evidence of clinically significant liver disease at the time of transplant readiness as determined by the clinical team
* Able to sign informed consent

Recipient Exclusion Criteria:

* Pregnant or nursing (lactating) women
* HBV positivity (Ag or DNA)
* Any contra-indication to kidney transplantation per center protocol

Donor Inclusion Criteria

* Detectable HCV NAT test
* KDPI score is less than ≤ 0.850
* Traditional Donor Selection Criteria Met - acceptable for transplantation per usual evaluation

Donor Exclusion Criteria

* Confirmed HIV
* Confirmed HBV positive (surface antigen or HBV DNA positive)
* Any standard contra-indication to donation noted in donor (significant malignancy, unusual infection, kidney anatomical damage or significant pathology)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-06-16 (Actual)

PRIMARY OUTCOMES:
Undetectable HCV RNA | 12 weeks post-treatment
  Negative HCV RNA 12 weeks after last dose of treatment
Rate of Serious and non-serious adverse events | 1 year post-transplant
  Determine safety of HCV+ to HCV- kidney transplantation by determining rate of adverse events related to HCV viremia or DAA treatment

IPD SHARING:
Plan to Share IPD: Yes
Anticipate to share coded data with collaborators
Supporting Information: Study Protocol
Time Frame: Ancicipate data would be available to share by 6 months are the final patient visit.
Access Criteria: Coded data would be shared with collaborators who have received IRB approval to use the data and have been approved by the PI for their collaboration.